CLINICAL TRIAL: NCT06190938
Title: The Relationship Between Diabetes, Its Neurological and Optical Complications, and Hearing Loss.
Brief Title: Diabetes Complications and Hearing Loss
Status: Completed | Type: Observational
Sponsor: Syrian Private University (Other)
Responsible Party: Principal Investigator, Mohamad Zaid Mohamad Samer Ahmad Abdalla, Dr in Damascus university in general internal medicine, Syrian Private University
Other Study IDs: Observation
Record Dates: First submitted 2023-10-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus; Diabetes Complications; Hearing Loss
Keywords: Diabetes retinopathy; Cataract
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Complications; Hearing Loss; Cataract

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The relation between diabetes, its neurological and optical complications with hearing loss

SUMMARY:
Observation study, shows the relation between diabetes, its neurological and optical complication and hearing loss, by asking participants questions about there age,BMI,job,the history of any cataract,diabetes retinopathy or heart attack,hypertension,swollen or tingling legs and take there consent to measure the hearing impairment.

ELIGIBILITY:
Inclusion Criteria:

* Diabetics who signed consent for the study.
* Diabetics who have filled out the form completely.
* Diabetics who have undergone a pure tone hearing screening test .

Exclusion Criteria:

* Patients with glandular disease causing hearing loss.
* Patients with traumatic ear injury.
* Patients who have recently had a middle or inner ear infection.
* History of acoustic neuroma.
* Patients are under active treatment with medications that have a toxic effect on the auditory cells.
* Patients with diabetic foot.
* The patient's occupation or residence is within a noisy environment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We collected participants from the clinical of Damascus hospital
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
The Demographic characteristics were classified into four groups: Gender, Financial status, Educational level, and Profession. | The study took 6 months to finish it with hard work, it was hard to reach our participants so it tooks 2 weeks from us for each participant to finish our survey
  Gender was either male or female. Income was divided into three categories: Low Income (those who were unable to provide even the basics for themselves), Fair Income (basics and some additional expenses), and High Income. Professions were divided into four types: Retired, Housewife, Worker and Student. Educational degree was categorized as Lower than High School, High School, or Higher than High School. Hypertension was measured and considered higher than normal when exceeded 140/90 mmHg. Both height and weight were measured to calculate the BMI of each subject.
  Weight was measured in kilograms. Height was measured in meters. BMI that scored less than 25, between 25-30, 30 or more was considered, underweight normal, and obese respectively.
  "The number of patients diagnosed with diabetes who showed signs of hearing impairment at certain stages of their lives, and how this related to other neurological signs, is being investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamad Zaid Ahmad Abdalla, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT06190938/Prot_SAP_000.pdf